CLINICAL TRIAL: NCT05552820
Title: Multicenter, Randomized, Single-blinded, Sham-Controlled Trial of Electroacupuncture on Mild-to-moderate Dry Eye
Brief Title: Electroacupuncture for Mild-to-moderate Dry Eye
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Shanghai Eye Disease Prevention and Treatment Center (Other); Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ShanghaiIAMM20220918
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye
Keywords: Dry eye; Electroacupuncture
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum Electroacupuncture (Experimental): Verum electroacupuncture treatment will be given 3 times a week, at least 1 day apart , for consecutive 4 weeks with a 24-week follow-up. Each session lasts for 30 min.
  Interventions: Device: Verum Electroacupuncture
- Sham Electroacupuncture (Sham Comparator): Sham electroacupuncture on non-acupoints plus non-penetrating plus no electrical stimulation will be given 3 times a week, at least 1 day apart , for consecutive 4 weeks with a 24-week follow-up. Each session lasts for 30 min.
  Interventions: Device: Sham Electroacupuncture

INTERVENTIONS:
Device: Verum Electroacupuncture — Acupoints: Cuanzhu (BL2), Taiyang (EX-HN5), Sibai (ST1), Sizhukong (TE23), Baihui (GV20), Fengchi (GB20), Hegu (LI4), Zusanli (ST36), Guangming (GB23), Sanyinjiao (SP6), and Taichong (LR3). All acupoints will be taken bilaterally, except Baihui (GV20). The subject is placed in the supine position with eyes close. After routine sterilization, the sterile polyethylene cylindrical needle pad will be adhered to the acupoints. Then, the sterile acupuncture needles (0.25 mm×0.40 mm, Hwato brand, China.) will be inserted into the skin through the needle pad. Twirling and lifting-thrusting manipulations will be performed on the acupoints until Deqi is reported by the subject. Two pairs of electrodes will be connected at the needle handles on BL2 and EX-HN5 with a 2 Hz, continuous-wave electro-stimulation provided by the electroacupuncture apparatus (SDZ-Ⅲ type, Hwato brand, China). The pulse amplitude is about 1-2 mA.
  Arms: Verum Electroacupuncture
Device: Sham Electroacupuncture — Sham acupoints: SA1(1 cm above BL2), SA2 (1 cm above SJ23)，SA3 (1 cm above EX-HN5), SA4 (1 cm lateral to ST2), SA5 (the midpoint of the line between GV20 and right EX-HN1), SA6 (the midpoint of the line between GB20 and SJ16), SA7 (1 cm lateral to LI4), SA8 (the midpoint of the line between ST36 and GB34), SA9 (the midpoint of the line between GB37 and BL58), SA10 (1 cm backward to SP6), SA11 (the midpoint of the line between LR3 and SP4). After routine sterilization, placebo needles will be used (Streitberger, Asia-med GmbH). The tingling sensation produced when the Streitberger needle is fixed on the skin causes the subject to believe that the needle is piercing the skin, simulating a skin puncture. The electric stimulator is applied to bilateral SA1 and SA3 with no current output. The exterior appearance, indicator light, prompt tone of the sham device, and stimulation parameters are all indistinguishable from the normal one.
  Arms: Sham Electroacupuncture

SUMMARY:
To determine if electroacupuncture acts as an dry eye treatment rather than a placebo, and identify if benefits are linked to corneal subbasal nerve changes and neuroimmunomodulatory indicators.

DETAILED DESCRIPTION:
Acupuncture is an important method in the treatment of diseases in Chinese medicine and plays an important role in the treatment of many diseases. Electroacupuncture (EA), as a combination of acupuncture and electric stimulation, is now widely used in research and clinical treatment. Our preliminary study found that compared with 0.1% sodium hyaluronate eye drops, EA exerted more beneficial and durable effects after four weeks of treatment. However, the placebo effect of EA cannot be ruled out yet. The aim of this study is to determine if EA acts as an dry eye treatment rather than a placebo, and identify if benefits are linked to corneal subbasal nerve changes.

This is a multicenter, randomized, subject-blinded, sham-controlled trial. A total of 168 participants with mild-to-moderate dry eye will be randomly assigned (1:1) to verum EA or non-penetrating non-acupoint sham EA (3 times weekly for 4 weeks), followed by a 24-week follow-up. The primary efficacy outcome is the change from baseline to week 4 in the Noninvasive Tear Breakup Time (NIBUT). Secondary efficacy outcomes include tear meniscus height (TMH), Schirmer I test (SⅠT), corneal topography, corneal and conjunctival sensation, scores of Ocular Surface Disease Index (OSDI), corneal fluorescein staining (CFS), Numerical rating scale (NRS), and Chinese Dry Eye Related Quality of Life Scale (CDERQOL) . Additionally, we will apply the Patient Health Questionnaire-9 (PHQ-9) and the Generalized Anxiety Disorder (GAD-7) to understand the mental health conditions of patients. IVCM will be performed to observe the morphological changes of the corneal basal nerve. The changes of NGF, CGRP, NPY, 8-OHDG, 4-HNE, MDA and other neuroimmunomodulatory indicators in tears and conjunctival cells will be detected by immunofluorescence, ELISA, or other techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the diagnostic criteria for dry eye according to the TFOS DEWS Ⅱ
* Ages 18-65 years, no gender limit

Exclusion Criteria:

* Diagnosed with severe dry eye
* Combined with other eye diseases (e.g. severe blepharitis, blepharospasm, conjunctival laxity, strabismus, amblyopia, glaucoma, cataract, fundus disease, ocular trauma)
* With active eye diseases or a history of eye surgery within 3 months
* Received acupuncture treatment or other dry eye treatment measures within 1 month that may influence the assessment of efficacy
* Previously experienced electroacupuncture intervention
* Pregnant or breastfeeding females
* Serious systemic diseases such as cardiovascular, cerebrovascular, hepatic, renal, and hematopoietic system and psychiatric disorders
* With autoimmune diseases such as Sjögren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, or ankylosing spondylitis
* With damaged, ulcerated, infected, or scarred skin at the selected acupoints
* Allergic to metal or tape

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Noninvasive Tear Breakup Time (NIBUT) | Baseline, Week 4, Week 8, Week 16, Week 28
  The interval between a complete blink and the first breakup of tear film (indicated by a break or deformed Placido disc image on the screen) will be recorded. The measurements are carried out 3 times and the average value is considered as NIBUT.

SECONDARY OUTCOMES:
Change From Baseline in Tear Meniscus Height (TMH) | Baseline, Week 4, Week 8, Week 16, Week 28
  The digital slit lamp (SL990N, CSO, Italy) is applied to take images of the tear meniscus at the lower lid margin in a dark room. The tear meniscus height directly below the central pupil is measured with the system's built-in caliper tool.
Change From Baseline in Ocular Surface Disease Index (OSDI) | Baseline, Week 4, Week 8, Week 16, Week 28
  The OSDI scale is used to assess subjective symptoms related to dry eye, including ocular symptoms, visual function and environmental triggers, with a total score ranging from 0 to 100. The higher the score, the more severe the subjective symptoms.
Change From Baseline in Corneal Fluorescein Staining (CFS) | Baseline, Week 4, Week 8, Week 16, Week 28
  Sodium fluorescein ophthalmic strips (Tianjin Jingming New Technology Development Co., Ltd., China) are used to evaluate corneal epithelial damage. According to the Oxford grading scheme, the CFS score ranges from 0 (no damage) to 5 (severe damage).
Change From Baseline in Corneal Topography | Baseline, Week 4, Week 8, Week 16, Week 28
  The corneal topography system is used to take photographs. The subjects are asked to blink naturally 3 to 4 times, and after the last full blink, they look at the central light source of the Placido disk for 10 s. The researchers take photographs of the anterior corneal surface immediately after the blink and at 10 s of continuous gaze. The SRI and SAI are systematically analyzed and obtained at 10 s.
Change From Baseline in Corneal and Conjunctival sensation | Baseline, Week 4, Week 8, Week 16, Week 28
  The Cochet-Bonnet perception meter (Luneau Chartres, France) will be used to evaluate the corneal perception (including central, superior, inferior, nasal, and temporal corneas, all 2 mm from the corneal rim) and conjunctival perception (including temporal and nasal bulbar conjunctivae, both 3 mm from the corneal rim; superior and inferior conjunctiva, at the center of the eyelid). The measured fiber length will be converted to g/mm2 according to the criteria provided by the supplier, with a higher threshold indicating a more insensitive perception.
Change From Baseline in Schirmer I test (SⅠT) | Baseline, Week 4, Week 8, Week 16, Week 28
  SⅠT will be performed using a tear detection filter strip (Tianjin Jingming New Technology Development Co., Ltd., China). Patients are requested to avoid eye movement. The strips will be removed after 5 min, and recorded the wetting length.
Change From Baseline in Numerical Rating Scale (NRS) | Baseline, Week 4, Week 8, Week 16, Week 28
  Subjects are asked to rate their current Iocular pain intensity in the right and left eye (0-10 numerical rating scale, NRS) followed by placement of 0.4% hydroxybuprocaine hydrochloride (Santen Pharmaceutical Co., LTD., Japan), and rerating of pain 30 seconds later.
Change From Baseline in Chinese Dry Eye Related Quality of Life Scale (CDERQOL) | Baseline, Week 4, Week 8, Week 16, Week 28
  CDERQOL includes 5 domians containing 45 items rated on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree).
Adverse events | Week 4
  Any adverse events will be recorded. EA-related adverse events include local bleeding, subcutaneous hematoma, pain, itch, infection, and generalized symptoms such as dizziness and palpitation during treatment.

OTHER OUTCOMES:
Change From Baseline in Generalized Anxiety Disorder (GAD-7) | Baseline, Week 4, Week 8, Week 16, Week 28
  The scale consists of 7 items with 4 frequency options for each question, ranging from "not at all (0)" to "almost every day (3)", with the following criteria: no anxiety (0-4); mild anxiety (5-9); moderate anxiety (10-14); and severe anxiety (15-21). 14 points); and severe anxiety (15-21 points).
Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) | Baseline, Week 4, Week 8, Week 16, Week 28
  The scale consists of 9 items with 4 frequency options for each question, ranging from "not at all (0)" to "almost every day (3)", with the following criteria: no depression (0-4); mild depression (5-9); moderate depression (10-14); moderate to severe depression (15-19); and severe depression (20-27). 14 points); moderate to severe depression (15-19 points); and severe depression (20-27 points)
Change in morphological changes of the corneal basal nerve | Baseline, Week 4
  In vivo confocal microscopy (IVCM) is performed to initially observe the morphological changes of the corneal basal nerve. IVCM images are taken with a Heidel-berg Retina Tomograph III (HRT III; Heidelberg Engi¬neering, Germany). The ACCMetrics analysis software (M.A. Dabbah, lmaging Science Biomedical Engineering, Manchester, UK) is used to calculate nerve morphological parameters for the selected images.
Change in neuroimmunomodulatory indicators in tears and conjunctival cells | Baseline, Week 4
  Schirmer test strip is s used to collect tears from patients before and after treatment. Conjunctival impression cytology is used to obtain conjunctival cells. Immunofluorescence, ELISA and other techniques are used to detect the changes in NGF, CGRP, NPY, 8-OHDG, 4-HNE, MDA and other neuroimmunomodulatory indicators in tears and conjunctival cells of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaopeng Ma, MD, PhD, Study Chair — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Guang Yang, Shanghai, China

REFERENCES:
- [Derived] Lu YQ, Yang G, Li MY, Hong J, Yang YT, Wang XJ, Kong XH, Zhao Y, Ma Z, Huang XY, Zou YL, Zhou XT, Ma XP. Electroacupuncture for mild-to-moderate dry eye: study protocol for a multicentre, randomised, single-blind, sham-controlled trial. BMJ Open. 2023 Dec 6;13(12):e069369. doi: 10.1136/bmjopen-2022-069369. PMID 38056935